CLINICAL TRIAL: NCT00708552
Title: Study AZ3110865, a Study Comparing SB-742457 or Donepezil Versus Placebo in Subjects With Mild-to-moderate Alzheimer's Disease
Brief Title: Study of SB-742457 or Donepezil Versus Placebo in Subjects With Mild-to-moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZ3110865
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Cognition; SB-742457
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- SB-742457 - 15mg (Experimental): SB-742457 - 15mg
  Interventions: Drug: SB-742457
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- SB-742457 - 35mg (Experimental): SB-742457 - 35mg
  Interventions: Drug: SB-742457
- Donepezil (Active Comparator)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: SB-742457 — investigational drug
  Arms: SB-742457 - 15mg; SB-742457 - 35mg
Drug: Donepezil — comparator
  Arms: Donepezil
Drug: Placebo — comparator
  Arms: Placebo

SUMMARY:
The study is designed to investigate the efficacy, safety and tolerability of SB-742457 versus placebo in subjects with mild-to-moderate Alzheimer's disease. SB-742457 is an experimental treatment which increases the levels of certain chemicals in the brain that are often decreased in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion criteria:

* Subjects and their caregivers must provide informed consent prior to study entry.
* Subjects must have a clinical diagnosis of probable mild-to-moderate Alzheimer's disease with a documented 6-month history of AD symptoms
* Subjects must have a regular caregiver who is willing to attend visits, oversee the subject's compliance with the study and report on the subject's status.
* Female subjects of child-bearing potential must agree to pregnancy testing and approved form of birth control.

Exclusion criteria:

* Diagnosis of possible, probable or definite vascular dementia.
* History/evidence of any other CNS disorder that could be interpreted as a cause of dementia
* History of known or suspected seizures, loss of consciousness or significant head trauma
* Subjects with ECG, blood pressure and laboratory values outside of protocol criteria are excluded.
* Subjects with known photosensitivity
* Subjects with a history of previous exposure to SB-742457, taking agents for which there is a theoretical risk of interaction with SB-742457, or taking medication for Alzheimer's disease or centrally acting agents which might impact study outcomes may not participate.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2008-07-04; Primary Completion 2010-03-01 (Actual); Study Completion 2010-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- Bulgaria (3):
  - GSK Investigational Site, Shumen
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Chile (3):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (20):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neuburg an der Donau, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Erbach im Odenwald, Hesse
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Siegen, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Hamburg
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Melíssia
  - GSK Investigational Site, Thessaloniki
- Mexico (5):
  - GSK Investigational Site, Aguascalientes, Ags, Aguascalientes
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Saltillo, Coahuila
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Mexico City
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Mosina
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Warsaw
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Africa (6):
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Loeventstein
  - GSK Investigational Site, Oakdale
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Rosebank
  - GSK Investigational Site, Sunninghill
- South Korea (2):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Seoul

REFERENCES:
- [Derived] Maher-Edwards G, Watson C, Ascher J, Barnett C, Boswell D, Davies J, Fernandez M, Kurz A, Zanetti O, Safirstein B, Schronen JP, Zvartau-Hind M, Gold M. Two randomized controlled trials of SB742457 in mild-to-moderate Alzheimer's disease. Alzheimers Dement (N Y). 2015 May 7;1(1):23-36. doi: 10.1016/j.trci.2015.04.001. eCollection 2015 Jun. PMID 29854923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 68 centers in the following 11 countries: Bulgaria, Chile, Czech Republic, Estonia, Germany, Greece, Korea, Mexico, Poland, Russia, and South Africa from 04 July 2008 to 09 Mar 2010 and a total of 967 participants were screened over the recruitment period of 55 weeks.
Pre-assignment Details: Of 967 participants screened, 618 (349 screen failures) entered into the placebo run-in period and a total of 576 (42 placebo run-in failures) were randomized of which 2 participants did not take study medication, formed Safety population (574) comprising of randomized participants who took atleast one dose of study medication.
Groups:
- Placebo: Participants received one tablet of matching placebo to SB-742457 (Week 1 to 4) and one capsule of matching placebo orally each evening just prior to going to bed (Week 4 to 24).
- SB-742457-15mg: Participants received one tablet of SB-742457-15 milligrams (mg) and one capsule of matching placebo to Donepezil orally each evening just prior to going to bed in the two treatment period (Week 1 to 4 and Week 4 to 24).
- SB-742457-35mg: Participants received one tablet of SB-742457-35 mg and one capsule of matching placebo to Donepezil orally each evening just prior to going to bed in the two treatment period (Week 1 to 4 and Week 4 to 24).
- Donepezil: Participants received Donepezil capsule by one-step titration 5mg Donepezil once daily (Week 1 to Week 4) before up-titrating at Visit 4 (Week 4) to 10 mg once daily dose for the remaining 20 weeks of the treatment period (Week 4 to 24) along with matching placebo to SB-747457.
Period: Overall Study
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Started | 145 | 145 | 133 | 151
Completed | 118 | 127 | 118 | 130
Not Completed | 27 | 18 | 15 | 21
Not completed — Adverse Event | 10 | 3 | 4 | 6
Not completed — Lack of Efficacy | 0 | 4 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 4 | 2 | 0 | 1
Not completed — Physician Decision | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 7 | 8 | 10

BASELINE CHARACTERISTICS:
Population: The population used to define the Baseline Characteristics was the Intent-to-Treat (ITT Population) which comprised of all participants randomized to treatment, and who received at least one dose of study medication and who had at least one post baseline assessment.
Groups:
- SB-742457-15mg: Participants received one tablet of SB-742457-15 mg and one capsule of matching placebo to Donepezil orally each evening just prior to going to bed in the two treatment period (Week 1 to 4 and Week 4 to 24).
- Total: Total of all reporting groups
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil | Total
Number analyzed (Participants) | 135 | 142 | 130 | 147 | 554
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.3 (6.80) | 72.4 (8.12) | 72.5 (7.38) | 71.1 (7.49) | 72.3 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 96 | 75 | 95 | 353
  Male | 48 | 46 | 55 | 52 | 201
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 9 | 5 | 9 | 26
  Asian | 4 | 7 | 6 | 6 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 3
  White | 128 | 126 | 118 | 130 | 502
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) Total Score at Week 24
Description: ADAS-Cog assesses a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items are evaluated by tests, but some are dependent on clinician ratings on a five point scale. The ADAS-Cog total score is the sum of the calculated scores for Questions 1 (Word recall task), 2 (Naming objects and fingers), and 7 (Word recognition task) and the scores recorded on the CRF for Questions 3 to 6 (Commands, Constructional praxis, Ideational praxis, Orientation) and 8 to 11 (Remembering test instructions, Spoken language ability, Word finding difficulty in spontaneous speech, Comprehension). The total score ranges from 0-70 with higher scores indicating greater dysfunction while lower indicates better cognitive function. Baseline was defined as the value at Week 0. Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 116 | 124 | 115 | 123
Score on scale | -0.3 (0.56) | 0.8 (0.58) | 0.4 (0.62) | -0.5 (0.45)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; ADAS-Cog Total Score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.159, Mixed model repeated measures; Mean Difference (Net) = 1.1, 95% CI 2-sided [-0.4 to 2.7]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; ADAS-Cog Total Score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.410, Mixed model repeated measures; Mean Difference (Net) = 0.7, 95% CI 2-sided [-0.9 to 2.3]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; ADAS-Cog Total Score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.821, Mixed model repeated measures; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.6 to 1.2]

2. Primary Outcome: Clinician's Interview-Based Impression of Change - Plus (CIBIC+) Score at Week 24
Description: The CIBIC+ is a rating scale derived from an interview with the participant and caregiver with an independent rater designed to measure several domains of participant function, such as mental/cognitive state, behavior, and functioning. The scores are rated on a scale of 1 to 7 as follows: 1 (marked improvement), 2 (moderately improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (moderately worse) and 7 (markedly worse).
Time Frame: Week 24
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 118 | 125 | 117 | 127
Score on scale | 4.0 (0.11) | 4.2 (0.10) | 3.9 (0.10) | 3.7 (0.10)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; CIBIC+ Score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.254, Mixed model repeated measures; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; CIBIC+ Score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.394, Mixed model repeated measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; CIBIC+ Score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.049, Mixed model repeated measures; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.6 to -0.0]

3. Secondary Outcome: Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Score at Week 24
Description: RBANS is an individually administered neurocognitive battery comprising 12 subtests across five domains (Attention, Language, Visuospatial/Constructional Abilities, and Immediate and Delayed memory). The scale is completed by a trained and experienced neurologist, psychiatrist or neuropsychologist, or another trained and experienced person. It is preferred that this individual is the same person who administers the ADAS-Cog, but he/she must be a separate individual from the person who completes the CIBIC+. The scale is based on the performance of the participant and takes approximately 25-30 minutes to administer. Raw total scores are calculated by adding up the scores for each of the 12 individual subtests and ranges between 0 and 311, where low score= (greater impairment) and high score=(better cognitive function). Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 116 | 125 | 115 | 127
Score on scale | -2.3 (1.44) | -4.0 (1.42) | -4.4 (1.49) | -0.3 (1.21)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; RBANS Total Score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.423, Mixed model repeated measures; Mean Difference (Net) = -1.6, 95% CI 2-sided [-5.6 to 2.3]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; RBANS Total Score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.305, Mixed model repeated measures; Mean Difference (Net) = -2.1, 95% CI 2-sided [-6.1 to 1.9]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; RBANS Total Score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.282, Mixed model repeated measures; Mean Difference (Net) = 2.0, 95% CI 2-sided [-1.7 to 5.7]

4. Secondary Outcome: Effect of Baseline Severity (Including Subgroup Analyses Based on Baseline Mini Mental State Examination [MMSE] Scores 16-26) on the Change From Baseline in ADAS-Cog Total Score, the Change From Baseline in RBANS Total Score at Week 24
Description: The MMSE was used to measure cognitive impairment. The MMSE consists of 11 tests namely orientation to time, orientation to place, registration, attention and calculation, recall, naming, repetition, comprehension, reading, writing and drawing corresponding to 5 domains orientation, memory, attention, and construction. All items were scored as 0 (incorrect response) or 1 (correct response). Total scores ranges from 0 to 30, with lower scores indicating greater cognitive impairment and higher scores indicating better function. Stratification by Baseline severity, using MMSE score at Baseline, with the strata being MMSE score of 10-15, 16-20 and 21-26. Two subgroups using MMSE score at Baseline were also examined, moderate 10-20 and mild 16-26. Data has been presented for participants with Baseline MMSE 16-26. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Intent-to-Treat (Baseline MMSE 16-26) which comprised of participants who had a baseline MMSE score of 16-26. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 99 | 110 | 98 | 113
Score on scale
  MMSE Score 16-26 on ADAS-Cog total score: number analyzed (Participants) | 88 | 99 | 86 | 94
  MMSE Score 16-26 on ADAS-Cog total score | -1.3 (0.55) | 0.1 (0.66) | -0.4 (0.73) | -1.0 (0.53)
  MMSE Score 16-26 on RBANS total score: number analyzed (Participants) | 87 | 100 | 85 | 95
  MMSE Score 16-26 on RBANS total score | -1.3 (1.61) | -2.4 (1.74) | -2.8 (1.82) | 1.1 (1.52)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 16-26 on ADAS-Cog Total score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.096, Mixed model repeated measures; Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.3 to 3.1]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 16-26 on ADAS-Cog Total score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.281, Mixed model repeated measures; Mean Difference (Net) = 1.0, 95% CI 2-sided [-0.8 to 2.8]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Baseline MMSE score of 16-26 on ADAS-Cog Total score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.630, Mixed model repeated measures; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.1 to 1.9]
Statistical Analysis 4: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 16-26 on RBANS Total score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.655, Mixed model repeated measures; Mean Difference (Net) = -1.1, 95% CI 2-sided [-5.7 to 3.6]
Statistical Analysis 5: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 16-26 on RBANS Total score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.545, Mixed model repeated measures; Mean Difference (Net) = -1.5, 95% CI 2-sided [-6.2 to 3.3]
Statistical Analysis 6: Comparison: Placebo vs Donepezil; Baseline MMSE score of 16-26 on RBANS Total score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.270, Mixed model repeated measures; Mean Difference (Net) = 2.4, 95% CI 2-sided [-1.9 to 6.8]

5. Secondary Outcome: Effect of Baseline Severity (Including Subgroup Analyses Based on Baseline [MMSE Scores 10-20) on the Change From Baseline in ADAS-Cog Total Score, the Change From Baseline in RBANS Total Score at Week 24
Description: The MMSE was used to measure cognitive impairment. The MMSE consists of 11 tests namely orientation to time, orientation to place, registration, attention and calculation, recall, naming, repetition, comprehension, reading, writing and drawing corresponding to 5 domains orientation, memory, attention, and construction. All items were scored as 0 (incorrect response) or 1 (correct response). Total scores ranges from 0 to 30, with lower scores indicating greater cognitive impairment and higher scores indicating better function. Stratification by Baseline severity, using MMSE score at Baseline, with the strata being MMSE score of 10-15, 16-20 and 21-26. Two subgroups using MMSE score at Baseline were also examined, moderate 10-20 and mild 16-26. Data has been presented for participants with Baseline MMSE 10-20. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Intent-to-Treat (Baseline MMSE 10-20) which comprised of participants who had a baseline MMSE score of 16-26. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 92 | 94 | 89 | 95
Score on scale
  MMSE Score 10-20 on ADAS-Cog total score: number analyzed (Participants) | 77 | 80 | 78 | 81
  MMSE Score 10-20 on ADAS-Cog total score | 0.0 (0.71) | 1.6 (0.76) | 1.3 (0.73) | -0.1 (0.58)
  MMSE Score 10-20 on RBANS total score: number analyzed (Participants) | 78 | 80 | 79 | 85
  MMSE Score 10-20 on RBANS total score | -3.7 (1.79) | -5.8 (1.73) | -4.8 (1.68) | -1.0 (1.44)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 10-20 on ADAS-Cog Total score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.138, Mixed model repeated measures; Mean Difference (Net) = 1.5, 95% CI 2-sided [-0.5 to 3.6]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 10-20 on ADAS-Cog Total score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.216, Mixed model repeated measures; Mean Difference (Net) = 1.3, 95% CI 2-sided [-0.7 to 3.2]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Baseline MMSE score of 10-20 on ADAS-Cog Total score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.921, Mixed model repeated measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.9 to 1.7]
Statistical Analysis 4: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 10-20 on RBANS Total score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.410, Mixed model repeated measures; Mean Difference (Net) = -2.1, 95% CI 2-sided [-7.0 to 2.9]
Statistical Analysis 5: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 10-20 on RBANS Total score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.667, Mixed model repeated measures; Mean Difference (Net) = -1.1, 95% CI 2-sided [-5.9 to 3.8]
Statistical Analysis 6: Comparison: Placebo vs Donepezil; Baseline MMSE score of 10-20 on RBANS Total score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.246, Mixed model repeated measures; Mean Difference (Net) = 2.7, 95% CI 2-sided [-1.9 to 7.2]

6. Secondary Outcome: Effect of Baseline Severity (Including Subgroup Analyses Based on Baseline MMSE Scores 16-26) on the CIBIC+ Score at Week 24
Description: The CIBIC+ is a rating scale derived from an interview with the participant and caregiver with an independent rater designed to measure several domains of participant function, such as mental/cognitive state, behavior, and functioning. The scores are rated on a scale of 1 to 7 as follows: 1 (marked improvement), 2 (moderately improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (moderately worse) and 7 (markedly worse). Stratification by Baseline severity, using MMSE score at Baseline, with the strata being MMSE score of 10-15, 16-20 and 21-26. Two subgroups using MMSE score at Baseline were also examined, moderate 10-20 and mild 16-26. Data has been presented for participants with Baseline MMSE 16-26. Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Intent-to-Treat (Baseline MMSE 16-26). Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 88 | 100 | 87 | 95
Score on scale | 3.8 (0.12) | 4.0 (0.12) | 3.7 (0.11) | 3.5 (0.11)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 16-26 on CBIC+ score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.146, Mixed model repeated measures; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 16-26 on CBIC+ score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.733, Mixed model repeated measures; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Baseline MMSE score of 16-26 on CBIC+ score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.145, Mixed model repeated measures; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

7. Secondary Outcome: Effect of Baseline Severity (Including Subgroup Analyses Based on Baseline MMSE Scores 10-20) on the CIBIC+ Score at Week 24
Description: The CIBIC+ is a rating scale derived from an interview with the participant and caregiver with an independent rater designed to measure several domains of participant function, such as mental/cognitive state, behavior, and functioning. The scores are rated on a scale of 1 to 7 as follows: 1 (marked improvement), 2 (moderately improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (moderately worse) and 7 (markedly worse). Higher scores indicate worst outcome. Stratification by Baseline severity, using MMSE score at Baseline, with the strata being MMSE score of 10-15, 16-20 and 21-26. Two subgroups using MMSE score at Baseline were also examined, moderate 10-20 and mild 16-26. Data has been presented for participants with baseline MMSE 10-20. Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Intent-to-Treat (Baseline MMSE 10-20). Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 79 | 80 | 80 | 85
Score on scale | 4.2 (0.15) | 4.4 (0.13) | 4.1 (0.12) | 3.9 (0.12)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 16-26 on CBIC+, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.295, Mixed model repeated measures; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 16-26 on CBIC+, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.495, Mixed model repeated measures; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Baseline MMSE score of 16-26 on CBIC+, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.166, Mixed model repeated measures; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.6 to 0.1]

8. Secondary Outcome: Change From Baseline in ADAS-Cog Total Score at Week 12
Description: ADAS-Cog assesses a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items are evaluated by tests, but some are dependent on clinician ratings on a five point scale. The ADAS-Cog total score is the sum of the calculated scores for Questions 1 (Word recall task), 2 (Naming objects and fingers), and 7 (Word recognition task) and the scores recorded on the CRF for Questions 3 to 6 (Commands, Constructional praxis, Ideational praxis, Orientation) and 8 to 11 (Remembering test instructions, Spoken language ability, Word finding difficulty in spontaneous speech, Comprehension). The total score ranges from 0-70 with higher scores indicating greater dysfunction while lower indicates better cognitive function. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 12.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 124 | 133 | 126 | 137
Score on scale | -0.1 (0.45) | 0.0 (0.46) | -0.2 (0.45) | -0.6 (0.40)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; ADAS-Cog Total Score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.847, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.1 to 1.4]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; ADAS-Cog Total Score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.833, Mixed Models Analysis; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.4 to 1.1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; ADAS-Cog Total Score, Placebo Vs Donepzil at Week 12; Test type: Superiority; p = 0.443, Mixed model repeated measures; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.6 to 0.7]

9. Secondary Outcome: CIBIC+ Score at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 126 | 133 | 126 | 139
Score on scale | 3.9 (0.08) | 4.0 (0.08) | 3.9 (0.09) | 3.7 (0.08)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; CIBIC+ Score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.320, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; CIBIC+ Score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.927, Mixed model repeated measures; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; CIBIC+ Score, Placebo Vs Donepzil at Week 12; Test type: Superiority; p = 0.059, Mixed model repeated measures; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.0]

10. Secondary Outcome: Change From Baseline in RBANS Total Score at Week 12
Description: RBANS is an individually administered neurocognitive battery comprising 12 subtests across five domains (Attention, Language, Visuospatial/Constructional Abilities, and Immediate and Delayed memory). The scale is completed by a trained and experienced neurologist, psychiatrist or neuropsychologist, or another trained and experienced person. It is preferred that this individual is the same person who administers the ADAS-Cog, but he/she must be a separate individual from the person who completes the CIBIC+. The scale is based on the performance of the participant and takes approximately 25-30 minutes to administer. Raw total scores are calculated by adding up the scores for each of the 12 individual subtests and ranges between 0 and 311, where low score= (greater impairment) and high score=(better cognitive function). Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 12.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 125 | 134 | 125 | 138
Score on scale | -6.7 (1.16) | -8.7 (1.24) | -5.9 (1.11) | -3.4 (1.06)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; RBANS total score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.257, Mixed model repeated measures; Mean Difference (Net) = -1.9, 95% CI 2-sided [-5.2 to 1.4]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; RBANS total score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.570, Mixed model repeated measures; Mean Difference (Net) = 0.9, 95% CI 2-sided [-2.2 to 4.0]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; RBANS total score, Placebo Vs Donepzil at Week 12; Test type: Superiority; p = 0.031, Mixed model repeated measures; Mean Difference (Net) = 3.4, 95% CI 2-sided [0.3 to 6.4]

11. Secondary Outcome: Effect of Baseline Severity (Including Subgroup Analyses Based on Baseline MMSE Scores 16-26) on the Change From Baseline in ADAS-Cog Total Score, the Change From Baseline in RBANS Total Score at Week 12
Description: The MMSE was used to measure cognitive impairment. The MMSE consists of 11 tests namely orientation to time, orientation to place, registration, attention and calculation, recall, naming, repetition, comprehension, reading, writing and drawing corresponding to 5 domains orientation, memory, attention, and construction. All items were scored as 0 (incorrect response) or 1 (correct response). Total scores ranges from 0 to 30, with lower scores indicating greater cognitive impairment and higher scores indicating better function. Stratification by Baseline severity, using MMSE score at Baseline, with the strata being MMSE score of 10-15, 16-20 and 21-26. Two subgroups using MMSE score at Baseline were also examined, moderate 10-20 and mild 16-26. Data has been presented for Participants with Baseline MMSE score 16-26. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 12.
Time Frame: Baseline (Week 0) and Week 12
Population: Intent-to-Treat (Baseline MMSE 16-26). Only those participants available at the specified time-points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 99 | 110 | 98 | 113
Score on scale
  MMSE Score 16-26 on ADAS-Cog total score: number analyzed (Participants) | 93 | 104 | 94 | 106
  MMSE Score 16-26 on ADAS-Cog total score | -0.6 (0.48) | -0.4 (0.47) | -0.5 (0.52) | -0.5 (0.42)
  MMSE Score 16-26 on RBANS total score: number analyzed (Participants) | 94 | 104 | 93 | 106
  MMSE Score 16-26 on RBANS total score | -7.5 (1.28) | -8.3 (1.51) | -4.4 (1.35) | -3.3 (1.31)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 16-26 on ADAS-Cog Total score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.798, Mixed model repeated measures; Mean Difference (Net) = 0.2, 95% CI 2-sided [-1.1 to 1.5]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 16-26 on ADAS-Cog Total score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.918, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.3 to 1.4]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Baseline MMSE score of 16-26 on ADAS-Cog Total score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.924, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.2 to 1.3]
Statistical Analysis 4: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 16-26 on RBANS Total score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.676, Mixed model repeated measures; Mean Difference (Net) = -0.8, 95% CI 2-sided [-4.7 to 3.0]
Statistical Analysis 5: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 16-26 on RBANS Total score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.086, Mixed model repeated measures; Mean Difference (Net) = 3.1, 95% CI 2-sided [-0.4 to 6.7]
Statistical Analysis 6: Comparison: Placebo vs Donepezil; Baseline MMSE score of 16-26 on RBANS Total score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.021, Mixed model repeated measures; Mean Difference (Net) = 4.2, 95% CI 2-sided [0.6 to 7.7]

12. Secondary Outcome: Effect of Baseline Severity (Including Subgroup Analyses Based on Baseline MMSE Scores 10-20) on the Change From Baseline in ADAS-Cog Total Score, the Change From Baseline in RBANS Total Score at Week 12
Description: The MMSE was used to measure cognitive impairment. The MMSE consists of 11 tests namely orientation to time, orientation to place, registration, attention and calculation, recall, naming, repetition, comprehension, reading, writing and drawing corresponding to 5 domains orientation, memory, attention, and construction. All items were scored as 0 (incorrect response) or 1 (correct response). Total scores ranges from 0 to 30, with lower scores indicating greater cognitive impairment and higher scores indicating better function. Stratification by Baseline severity, using MMSE score at Baseline, with the strata being MMSE score of 10-15, 16-20 and 21-26. Two subgroups using MMSE score at Baseline were also examined, moderate 10-20 and mild 16-26. Data has been presented for participants with Baseline MMSE score 10-20. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 12.
Time Frame: Baseline (Week 0) and Week 12
Population: Intent-to-Treat (Baseline MMSE 10-20). Only those participants available at the specified time-points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 92 | 94 | 89 | 95
Score on scale
  MMSE Score 10-20 on ADAS-Cog total score: number analyzed (Participants) | 85 | 88 | 87 | 88
  MMSE Score 10-20 on ADAS-Cog total score | 0.4 (0.51) | 0.4 (0.61) | 0.2 (0.60) | -0.9 (0.51)
  MMSE Score 10-20 on RBANS total score: number analyzed (Participants) | 85 | 89 | 87 | 89
  MMSE Score 10-20 on RBANS total score | -6.4 (1.36) | -10.0 (1.29) | -6.8 (1.26) | -1.7 (1.20)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 10-20 on ADAS-Cog Total score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.908, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.5 to 1.7]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 10-20 on ADAS-Cog Total score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.826, Mixed model repeated measures; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.7 to 1.4]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Baseline MMSE score of 10-20 on ADAS-Cog Total score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.088, Mixed model repeated measures; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.7 to 0.2]
Statistical Analysis 4: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 10-20 on RBANS Total score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.053, Mixed model repeated measures; Mean Difference (Net) = -3.6, 95% CI 2-sided [-7.3 to 0.0]
Statistical Analysis 5: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 10-20 on RBANS Total score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.848, Mixed Models Analysis; Mean Difference (Net) = -0.4, 95% CI 2-sided [-4.0 to 3.3]
Statistical Analysis 6: Comparison: Placebo vs Donepezil; Baseline MMSE score of 10-20 on RBANS Total score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.011, Mixed model repeated measures; Mean Difference (Net) = 4.7, 95% CI 2-sided [1.1 to 8.2]

13. Secondary Outcome: Effect of Baseline Severity (Including Subgroup Analyses Based on Baseline MMSE Scores 16-26) on the CIBIC+ Score at Week 12
Description: The CIBIC+ is a rating scale derived from an interview with the participant and caregiver with an independent rater designed to measure several domains of participant function, such as mental/cognitive state, behavior, and functioning. The scores are rated on a scale of 1 to 7 as follows: 1 (marked improvement), 2 (moderately improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (moderately worse) and 7 (markedly worse). Stratification by Baseline severity, using MMSE score at Baseline, with the strata being MMSE score of 10-15, 16-20 and 21-26. Two subgroups using MMSE score at Baseline were also examined, moderate 10-20 and mild 16-26. Data has been presented for participants with Baseline MMSE score 16-26.
Time Frame: Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 94 | 104 | 94 | 107
Score on scale | 3.8 (0.08) | 3.8 (0.09) | 3.7 (0.10) | 3.6 (0.08)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 16-26 on CIBIC+ score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.671, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 16-26 on CIBIC+ Total score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.413, Mixed model repeated measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Baseline MMSE score of 16-26 on CIBIC+ Total score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.245, Mixed model repeated measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.1]

14. Secondary Outcome: Effect of Baseline Severity (Including Subgroup Analyses Based on Baseline MMSE Scores 10-20) on the CIBIC+ Score at Week 12
Description: The CIBIC+ is a rating scale derived from an interview with the participant and caregiver with an independent rater designed to measure several domains of participant function, such as mental/cognitive state, behavior, and functioning. The scores are rated on a scale of 1 to 7 as follows: 1 (marked improvement), 2 (moderately improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (moderately worse) and 7 (markedly worse). Stratification by Baseline severity, using MMSE score at Baseline, with the strata being MMSE score of 10-15, 16-20 and 21-26. Two subgroups using MMSE score at Baseline were also examined, moderate 10-20 and mild 16-26. Data has been presented for participants with Baseline MMSE score 10-20.
Time Frame: Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 86 | 88 | 87 | 90
Score on scale | 4.0 (0.10) | 4.1 (0.10) | 4.1 (0.11) | 3.7 (0.11)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Baseline MMSE score of 10-20 on CIBIC+ score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.369, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Baseline MMSE score of 10-20 on CIBIC+ Total score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.550, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Baseline MMSE score of 10-20 on CIBIC+ Total score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.082, Mixed model repeated measures; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.5 to 0.0]

15. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) Total Score at Weeks 12 and 24
Description: The ADCS-ADL measures functional impairment in terms of activities of daily living. The ADCS-ADL is an interviewer-administered informant-based scale where the informant (caregiver) responds to 23 activities of daily living questions (i.e. those necessary for personal care, communicating and interacting with other people, maintaining a household, conducting hobbies and interests, making judgments and decisions) about the participant. The questions range from basic to instrumental activities of daily living and take approximately 20 minutes to complete. The Total score ranges from 0-78 and a higher score signifies greater functional ability and lower scores indicating greater impairment. The total score is the sum of all items and sub-questions. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Weeks 12 and 24.
Time Frame: Baseline (Week 0) and Weeks 12 and 24
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 135 | 142 | 130 | 147
Score on scale
  ADCS-ADL Total score at Week 12: number analyzed (Participants) | 126 | 133 | 124 | 139
  ADCS-ADL Total score at Week 12 | -0.4 (0.59) | -1.1 (0.65) | -0.1 (0.64) | 0.2 (0.62)
  ADCS-ADL Total score at Week 24: number analyzed (Participants) | 118 | 123 | 114 | 128
  ADCS-ADL Total score at Week 24 | -1.0 (0.71) | -1.4 (0.68) | -1.1 (0.81) | -1.2 (0.82)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; ADCS-ADL Total score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.417, Mixed model repeated measures; Mean Difference (Net) = -0.7, 95% CI 2-sided [-2.4 to 1.0]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; ADCS-ADL Total score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.725, Mixed model repeated measures; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.4 to 2.0]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; ADCS-ADL Total score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.506, Mixed model repeated measures; Mean Difference (Net) = 0.6, 95% CI 2-sided [-1.1 to 2.2]
Statistical Analysis 4: Comparison: Placebo vs SB-742457-15mg; ADCS-ADL Total score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.723, Mixed model repeated measures; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.3 to 1.6]
Statistical Analysis 5: Comparison: Placebo vs SB-742457-35mg; ADCS-ADL Total score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.919, Mixed model repeated measures; Median Difference (Net) = -0.1, 95% CI 2-sided [-2.2 to 2.0]
Statistical Analysis 6: Comparison: Placebo vs Donepezil; ADCS-ADL Total score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.896, Mixed model repeated measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-2.3 to 2.0]

16. Secondary Outcome: Change From Baseline in Cornell Scale for Depression in Dementia (CSDD) Total Score at Week 24
Description: The CSDD is used to assess signs and symptoms of major depression in demented participants. The CSDD scale contains 19 items on mood-related signs of depression, behavioral disturbance, physical signs of depression, cyclic functions and ideational disturbances, where each item is rated for severity on a scale of 0-2 (0=absent, 1=mild/intermittent, 2=severe). Scores above 10 (probable major depression),scores above 18 (definite major depression), scores below 6 (absence of significant depressive symptoms). The total score was calculated as a weighted average of the scores provided for the remaining 18 questions as follows: Imputed Total= Observed Total Score x 1+ Maximum Score of the missing value/ Sum of the Maximum Score of the non -missing values) and ranges from 0-38. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 118 | 125 | 117 | 128
Score on scale | 0.0 (0.26) | -0.1 (0.25) | 0.3 (0.26) | 0.3 (0.25)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; CSDD Total score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.594, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.9 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; CSDD Total score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.523, ANCOVA; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.5 to 0.9]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; CSDD Total score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.429, ANCOVA; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.4 to 1.0]

17. Secondary Outcome: Change From Baseline in MMSE Total Score at Week 24
Description: The MMSE is used to test for cognitive dysfunction. The scale is completed by a trained and experienced neurologist/psychiatrist/neuropsychologist based on the performance of the participants, and takes approximately 5 to 10 minutes to administer. It consists of 11 tests namely orientation to time, orientation to place, registration, attention and calculation, recall, naming, repetition, comprehension, reading, writing, drawing across 5 sections (orientation, registration, attention-calculation, recall, and language). Scoring was done by circling 0 if the response was incorrect, or 1 if the response was correct. Scores range from 0 to 30, with lower scores indicating greater cognitive impairment and higher scores indicating better cognitive function. The total MMSE score was a sum of all item scores. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 118 | 124 | 117 | 128
Score on scale | -0.3 (0.29) | -0.3 (0.28) | -0.1 (0.29) | 0.5 (0.27)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; MMSE Total score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.966, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.8 to 0.8]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; MMSE Total score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.505, ANCOVA; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.5 to 1.1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; MMSE Total score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.044, ANCOVA; Mean Difference (Net) = 0.8, 95% CI 2-sided [0.0 to 1.6]

18. Secondary Outcome: Change From Baseline in ADCS-ADL-Basic Score; ADCS-ADL: Instrumental Score and ADCS-ADL: Total Independence Score at Weeks 12 and 24
Description: Basic score was calculated as the sum of questions 1-6b and ranges from 0-22 (activities included are: eating, walking, using the toilet, bathing, grooming and dressing) and Instrumental score, sum of questions 7-23, ranges from 0-56 (activities included are: using the telephone, watching television, conversations, clearing dishes, personal belongings, making drinks, making snacks, taking rubbish out, getting out and about, shopping, keeping appointments, being left alone, current events, reading, writing, pastimes/hobbies, household chores). Total independence score is calculated by re-scoring the individual questions for each activity. The total independence score therefore ranges between 0 to 23, where 23 indicates that a participant is independent (based on these 23 ADL). Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Weeks 12 and 24.
Time Frame: Baseline (Week 0) and Weeks 12 and 24
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 135 | 142 | 130 | 147
Score on scale
  Basic score at Week 12: number analyzed (Participants) | 126 | 133 | 124 | 139
  Basic score at Week 12 | -0.6 (0.17) | -0.5 (0.19) | -0.4 (0.24) | -0.2 (0.17)
  Basic score at Week 24: number analyzed (Participants) | 118 | 123 | 114 | 128
  Basic score at Week 24 | -0.7 (0.20) | -0.7 (0.19) | -0.6 (0.24) | -0.8 (0.23)
  Instrumental score at Week 12: number analyzed (Participants) | 126 | 133 | 124 | 139
  Instrumental score at Week 12 | 0.2 (0.50) | -0.6 (0.55) | 0.3 (0.52) | 0.4 (0.55)
  Instrumental score at Week 24: number analyzed (Participants) | 118 | 124 | 114 | 128
  Instrumental score at Week 24 | -0.3 (0.60) | -0.7 (0.61) | -0.5 (0.68) | -0.4 (0.70)
  Total Independence Score at Week 12: number analyzed (Participants) | 126 | 133 | 124 | 139
  Total Independence Score at Week 12 | -0.1 (0.23) | -0.1 (0.23) | 0.2 (0.24) | 0.2 (0.23)
  Total Independence Score at Week 24: number analyzed (Participants) | 118 | 124 | 114 | 128
  Total Independence Score at Week 24 | -0.3 (0.27) | -0.2 (0.26) | -0.1 (0.29) | -0.1 (0.30)
Statistical Analysis 1: Comparison: Placebo vs SB-742457-15mg; Basic Score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.869, Mixed model repeated measures; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs SB-742457-35mg; Basic Score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.500, Mixed model repeated measures; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.4 to 0.8]
Statistical Analysis 3: Comparison: Placebo vs Donepezil; Basic Score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.140, Mixed model repeated measures; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.1 to 0.8]
Statistical Analysis 4: Comparison: Placebo vs SB-742457-15mg; Basic Score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.910, Mixed model repeated measures; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.6 to 0.5]
Statistical Analysis 5: Comparison: Placebo vs SB-742457-35mg; Basic Score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.774, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 6: Comparison: Placebo vs Donepezil; Basic Score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.726, Mixed model repeated measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.7 to 0.5]
Statistical Analysis 7: Comparison: Placebo vs SB-742457-15mg; Instrumental Score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.292, Mixed model repeated measures; Mean Difference (Net) = -0.8, 95% CI 2-sided [-2.2 to 0.7]
Statistical Analysis 8: Comparison: Placebo vs SB-742457-35mg; Instrumental Score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.946, Mixed model repeated measures; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.3 to 1.4]
Statistical Analysis 9: Comparison: Placebo vs Donepezil; Instrumental Score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.802, Mixed model repeated measures; Mean Difference (Net) = 0.2, 95% CI 2-sided [-1.3 to 1.6]
Statistical Analysis 10: Comparison: Placebo vs SB-742457-15mg; Instrumental Score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.636, Mixed model repeated measures; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.1 to 1.3]
Statistical Analysis 11: Comparison: Placebo vs SB-742457-35mg; Instrumental Score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.752, Mixed model repeated measures; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.0 to 1.5]
Statistical Analysis 12: Comparison: Placebo vs Donepezil; Instrumental Score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.920, Mixed model repeated measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.9 to 1.7]
Statistical Analysis 13: Comparison: Placebo vs SB-742457-15mg; Total Independence Score, Placebo Vs SB-742457-15mg at Week 12; Test type: Superiority; p = 0.972, Mixed model repeated measures; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 14: Comparison: Placebo vs SB-742457-35mg; Total Independence Score, Placebo Vs SB-742457-35mg at Week 12; Test type: Superiority; p = 0.378, Mixed model repeated measures; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.4 to 0.9]
Statistical Analysis 15: Comparison: Placebo vs Donepezil; Total Independence Score, Placebo Vs Donepezil at Week 12; Test type: Superiority; p = 0.346, Mixed model repeated measures; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.3 to 0.9]
Statistical Analysis 16: Comparison: Placebo vs SB-742457-15mg; Total Independence Score, Placebo Vs SB-742457-15mg at Week 24; Test type: Superiority; p = 0.720, Mixed model repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.6 to 0.9]
Statistical Analysis 17: Comparison: Placebo vs SB-742457-35mg; Total Independence Score, Placebo Vs SB-742457-35mg at Week 24; Test type: Superiority; p = 0.598, Mixed model repeated measures; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.6 to 1.0]
Statistical Analysis 18: Comparison: Placebo vs Donepezil; Total Independence Score, Placebo Vs Donepezil at Week 24; Test type: Superiority; p = 0.480, Mixed model repeated measures; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.5 to 1.1]

19. Secondary Outcome: Number of Participants With Any Adverse Event (Serious and Non-serious) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury. Number of participants with any adverse event (serious and non-serious) and SAEs were reported.
Time Frame: Upto Week 24
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 145 | 145 | 133 | 151
Participants
  Any AE | 45 | 42 | 39 | 65
  Any SAE | 7 | 7 | 3 | 10

20. Secondary Outcome: Number of Participants With Vital Signs Data of Potential Clinical Concern (PCC) Any Time on Treatment (ATOT)
Description: Vital sign measurements included systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Heart Rate (HR), Body weight (BW). SBP and DBP and HR were measured once after the participant sat quietly for at least 5 minutes and in addition, upon standing to assess participants for postural hypotension. DBP was measured at the disappearance of Korotkoff sounds (Phase V). The plethysmographic method (preferably with a column sphygmomanometer where available) was used to measure blood pressure throughout the study. Body weight was measured, without shoes and wearing light clothing. The PCC range were as follows: SBP (Reference Range [RR] <90-140> Increase from Baseline [IFB]>=40 and decrease from baseline [DFB] >=30), DBP (RR < 50-90> IFB>=30 and DFB >=20), HR (RR <50-100> IFB >=30 and DFB >=30, BW (IFB >= 7% and DFB >=7%).
Time Frame: Upto Week 24
Population: Safety population. Only those participants with data available at the indicated time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 140 | 143 | 133 | 149
Participants
  SBP sitting ATOT <90 or > 140 and IFB >=40 | 1 | 2 | 2 | 0
  SBP standing ATOT <90 or > 140 and IFB >=40 | 0 | 3 | 3 | 1
  SBP standing ATOT <90 or > 140 and DFB >=30 | 0 | 0 | 0 | 4
  SBP orthostatic, fall in SBP >30 | 0 | 0 | 3 | 1
  DBP sitting ATOT <50 or > 90 and IFB >=30 | 0 | 0 | 1 | 1
  DBP sitting ATOT <50 or > 90 and DFB >=20 | 0 | 1 | 0 | 0
  DBP standing ATOT <50 or > 90 and IFB >=30 | 2 | 0 | 2 | 0
  DBP standing ATOT <50 or > 90 and DFB >=20 | 0 | 0 | 0 | 1
  DBP orthostatic, fall in SBP >20 | 0 | 0 | 1 | 1
  HR sitting ATOT <50 or >100 and DFB >=30 | 0 | 1 | 0 | 0
  HR standing ATOT <50 or >100 and IFB >=30 | 1 | 0 | 0 | 0
  HR orthostatic, increase in HR>= >20 | 5 | 2 | 2 | 6
  Weight, IFB>=7% | 4 | 4 | 6 | 6
  Weight, DFB>=7% | 6 | 8 | 5 | 10

21. Secondary Outcome: Number of Participants With Hematology Data of PCC ATOT
Description: Hematology parameters included hematocrit ratio (reference range males 0.410-0.500, females 0.350-0.460 [18-64 years] and males 0.360-0.490, females 0.330-0.460 [65+ years]), hemoglobin grams per liter (13.8-17.2), lymphocytes giga per liter (0.85-4.10), monocytes giga per liter (0.20-1.10), platelet count giga per liter (130-400), segmented neutrophils giga per liter (1.80-8.00), total neutrophils (1.80-8.00). Data has been presented in a consolidated format for hematology parameters high and low from the reference range of PCC ATOT.
Time Frame: Upto Week 24
Population: Safety population. Only those participants available at the specified time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 145 | 145 | 133 | 151
Participants
  Hematocrit, ATOT, low: number analyzed (Participants) | 138 | 143 | 132 | 149
  Hematocrit, ATOT, low | 1 | 0 | 0 | 1
  Hemoglobin, ATOT. low: number analyzed (Participants) | 138 | 143 | 132 | 149
  Hemoglobin, ATOT. low | 2 | 1 | 2 | 6
  Lymphocytes, ATOT, low: number analyzed (Participants) | 138 | 143 | 132 | 149
  Lymphocytes, ATOT, low | 4 | 5 | 3 | 2
  Lymphocytes, ATOT, high: number analyzed (Participants) | 138 | 143 | 132 | 149
  Lymphocytes, ATOT, high | 0 | 2 | 0 | 0
  Monocytes, ATOT, low: number analyzed (Participants) | 138 | 143 | 132 | 149
  Monocytes, ATOT, low | 17 | 10 | 9 | 24
  Platelet count, ATOT, low: number analyzed (Participants) | 138 | 143 | 131 | 149
  Platelet count, ATOT, low | 3 | 2 | 2 | 2
  Segmented neutrophils, ATOT, low: number analyzed (Participants) | 138 | 143 | 132 | 149
  Segmented neutrophils, ATOT, low | 2 | 1 | 0 | 1
  Segmented neutrophils, ATOT, high: number analyzed (Participants) | 138 | 143 | 132 | 149
  Segmented neutrophils, ATOT, high | 1 | 1 | 1 | 1
  Total neutrophils, ATOT, low: number analyzed (Participants) | 138 | 143 | 132 | 149
  Total neutrophils, ATOT, low | 2 | 1 | 0 | 1
  Total neutrophils, ATOT, high: number analyzed (Participants) | 138 | 143 | 132 | 149
  Total neutrophils, ATOT, high | 0 | 1 | 1 | 1
  White blood cell count, ATOT, low: number analyzed (Participants) | 138 | 143 | 132 | 149
  White blood cell count, ATOT, low | 2 | 0 | 1 | 1
  White blood cell count, ATOT, high: number analyzed (Participants) | 138 | 143 | 132 | 149
  White blood cell count, ATOT, high | 0 | 3 | 1 | 1

22. Secondary Outcome: Number of Participants With Chemistry Data of PCC ATOT
Description: Clinical chemistry parameters included alanine amino transferase international units per liter (IU/L) RR [0-48], alkaline phosphatase IU/L (20-125), aspartate amino transferase international units per liter (0-55), blood urea nitrogen/creatinine ratio (24-101), calcium millimoles per liter (mmol/L) [2.12-2.56], carbon dioxide content/bicarbonate mmol/L (20-32), cholesterol mmol/L (0.00-5.15), creatine kinase IU/L (males 0-235 and females 0-190), creatinine micromoles per liter (umol/L) [44-124], direct bilirubin umol/L (0-6), gamma glutamyl transferase IU/L (males 0-65 and females 0-45), glucose mmol/L (3.9-6.9), low density lipoprotein cholesterol mmol/L (0.00-3.35), lactate dehydrogenase IU/L (0-270), potassium mmol/L (3.5-5.3), sodium mmol/L (135-146), total bilirubin umol/L (0-22), triglycerides mmol/L (0.00-2.24), urea/blood urea nitrogen mmol/L (2.5-10.5). Data has been presented in a consolidated format for clinical chemistry parameters high and low from the RR of PCC ATOT.
Time Frame: Upto Week 24
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 145 | 145 | 133 | 151
Participants
  Alanine Amino Transferase, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Alanine Amino Transferase, ATOT, high | 2 | 0 | 0 | 1
  Alkaline Phosphatase, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Alkaline Phosphatase, ATOT, high | 1 | 0 | 2 | 6
  Aspartate Amino Transferase, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Aspartate Amino Transferase, ATOT, high | 0 | 0 | 0 | 1
  Blood urea nitrogen/Creatinine ratio, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Blood urea nitrogen/Creatinine ratio, ATOT, high | 1 | 4 | 0 | 3
  Calcium, ATOT, low: number analyzed (Participants) | 138 | 142 | 132 | 149
  Calcium, ATOT, low | 0 | 0 | 1 | 0
  Carbon dioxide content/Bicarbonate, ATOT, low: number analyzed (Participants) | 138 | 142 | 132 | 149
  Carbon dioxide content/Bicarbonate, ATOT, low | 1 | 0 | 0 | 0
  Cholesterol, ATOT, high: number analyzed (Participants) | 120 | 126 | 118 | 134
  Cholesterol, ATOT, high | 5 | 5 | 2 | 7
  Creatine Kinase, ATOT, high: number analyzed (Participants) | 120 | 126 | 118 | 134
  Creatine Kinase, ATOT, high | 3 | 1 | 5 | 7
  Creatinine, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Creatinine, ATOT, high | 3 | 1 | 4 | 1
  Direct Bilirubin, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Direct Bilirubin, ATOT, high | 0 | 0 | 0 | 1
  Gamma Glutamyl Transferase, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Gamma Glutamyl Transferase, ATOT, high | 3 | 1 | 4 | 4
  Glucose, ATOT, low: number analyzed (Participants) | 138 | 142 | 132 | 149
  Glucose, ATOT, low | 7 | 5 | 8 | 6
  Glucose, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Glucose, ATOT, high | 27 | 16 | 23 | 22
  Low Density Lipoprotein Cholesterol, ATOT, high: number analyzed (Participants) | 117 | 126 | 117 | 132
  Low Density Lipoprotein Cholesterol, ATOT, high | 21 | 26 | 12 | 25
  Lactate Dehydrogenase, ATOT, high: number analyzed (Participants) | 120 | 126 | 118 | 134
  Lactate Dehydrogenase, ATOT, high | 0 | 1 | 0 | 0
  Potassium, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Potassium, ATOT, high | 5 | 5 | 2 | 7
  Sodium, ATOT, low: number analyzed (Participants) | 138 | 142 | 132 | 149
  Sodium, ATOT, low | 0 | 2 | 0 | 0
  Sodium, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Sodium, ATOT, high | 0 | 0 | 0 | 1
  Total Bilirubin, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Total Bilirubin, ATOT, high | 1 | 1 | 0 | 2
  Triglycerides, ATOT, high: number analyzed (Participants) | 120 | 126 | 118 | 134
  Triglycerides, ATOT, high | 0 | 0 | 0 | 1
  Urea/Blood urea nitrogen, ATOT, high: number analyzed (Participants) | 138 | 142 | 132 | 149
  Urea/Blood urea nitrogen, ATOT, high | 7 | 6 | 8 | 4

23. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Alanine Amino Transferase, Alkaline Phosphatase, Aspartate Amino Transferase, Creatine Kinase, Gamma Glutamyl Transferase and Lactate Dehydrogenase at Week 24
Description: Clinical chemistry parameters included alanine amino transferase, alkaline phosphatase, aspartate amino transferase, creatine kinase, gamma glutamyl transferase and lactate dehydrogenase. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Weeks 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 145 | 145 | 133 | 151
IU/L
  Alanine amino transferase at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Alanine amino transferase at Week 24 | -0.3 (8.76) | 0.0 (4.88) | -0.1 (6.77) | 1.6 (29.47)
  Alkaline phosphatase at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Alkaline phosphatase at Week 24 | -3.4 (15.71) | -0.1 (10.91) | 0.8 (14.63) | 2.0 (17.81)
  Aspartate amino transferase at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Aspartate amino transferase at Week 24 | -0.3 (6.15) | 0.0 (3.80) | -0.1 (6.88) | 0.5 (12.88)
  Creatine kinase at Week 24: number analyzed (Participants) | 111 | 117 | 115 | 126
  Creatine kinase at Week 24 | -16.8 (242.93) | -5.4 (47.97) | 16.2 (157.67) | 0.6 (82.86)
  Gamma glutamyl transferase at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Gamma glutamyl transferase at Week 24 | -1.5 (13.06) | -0.2 (11.23) | -1.3 (15.08) | 3.6 (32.97)
  Lactate dehydrogenase at Week 24: number analyzed (Participants) | 111 | 117 | 115 | 126
  Lactate dehydrogenase at Week 24 | 0.8 (25.09) | -2.9 (28.88) | -0.4 (22.65) | -1.2 (25.99)

24. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Albumin and Total Protein at Week 24
Description: Clinical chemistry parameters included albumin and total protein. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 111 | 117 | 115 | 126
grams per liter
  Albumin at Week 24 | -0.5 (2.37) | -0.5 (2.44) | -0.6 (2.54) | -0.8 (2.62)
  Total protein at Week 24 | -0.8 (3.52) | -0.9 (4.00) | -1.3 (3.50) | -1.2 (3.62)

25. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter Blood Urea Nitrogen /Creatinine Ratio at Week 24
Description: Clinical chemistry parameter included blood urea nitrogen /creatinine ratio. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 115 | 121 | 116 | 127
Ratio | 0.8 (19.99) | 2.3 (19.32) | -3.7 (17.44) | -0.3 (17.76)

26. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Calcium, CO2 Content/Bicarbonate, Chloride, Glucose, HDL Cholesterol, LDL Cholesterol, Magnesium, Phosphorus, Potassium, Sodium, Triglycerides, Urea/Blood Urea Nitrogen at Week 24
Description: Clinical chemistry parameters included calcium, CO2 content/bicarbonate, chloride, glucose, HDL cholesterol, LDL cholesterol, magnesium, phosphorus, potassium, sodium, triglycerides, urea/blood urea nitrogen. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 145 | 145 | 133 | 151
mmol/L
  Calcium at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Calcium at Week 24 | -0.008 (0.0910) | -0.012 (0.0956) | -0.025 (0.1215) | -0.013 (0.0932)
  CO2 content/bicarbonate at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  CO2 content/bicarbonate at Week 24 | 0.5 (2.91) | 0.3 (2.46) | -0.5 (3.01) | 0.5 (2.84)
  Chloride at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Chloride at Week 24 | 0.2 (2.54) | 0.3 (2.97) | 0.1 (2.87) | -0.0 (2.70)
  Glucose at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Glucose at Week 24 | 0.02 (1.108) | 0.03 (1.327) | 0.14 (1.808) | 0.07 (1.605)
  HDL cholesterol at Week 24: number analyzed (Participants) | 111 | 117 | 115 | 126
  HDL cholesterol at Week 24 | -0.023 (0.2272) | -0.060 (0.2402) | -0.060 (0.3050) | -0.035 (0.2477)
  LDL cholesterol at Week 24: number analyzed (Participants) | 107 | 116 | 113 | 122
  LDL cholesterol at Week 24 | 0.149 (0.8387) | -0.032 (0.6176) | -0.115 (0.5971) | -0.032 (0.7417)
  Magnesium at Week 24: number analyzed (Participants) | 111 | 117 | 115 | 126
  Magnesium at Week 24 | -0.001 (0.0606) | -0.007 (0.0538) | -0.002 (0.0569) | -0.001 (0.0591)
  Phosphorus at Week 24: number analyzed (Participants) | 111 | 117 | 115 | 126
  Phosphorus at Week 24 | 0.010 (0.1435) | -0.018 (0.1529) | 0.043 (0.1728) | 0.026 (0.1752)
  Potassium at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Potassium at Week 24 | -0.00 (0.450) | 0.09 (0.458) | 0.04 (0.440) | 0.05 (0.450)
  Sodium at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Sodium at Week 24 | 0.1 (2.24) | 0.0 (2.57) | -0.2 (2.43) | 0.4 (2.31)
  Triglycerides at Week 24: number analyzed (Participants) | 111 | 117 | 115 | 126
  Triglycerides at Week 24 | -0.040 (0.8750) | -0.071 (0.7146) | -0.024 (0.7678) | 0.082 (1.0874)
  Urea/blood urea nitrogen at Week 24: number analyzed (Participants) | 115 | 121 | 116 | 127
  Urea/blood urea nitrogen at Week 24 | 0.06 (1.642) | 0.29 (1.510) | 0.14 (1.467) | 0.10 (1.453)

27. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Creatinine, Direct Bilirubin and Total Bilirubin at Week 24
Description: Clinical chemistry parameters included creatinine, direct bilirubin and total bilirubin. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 115 | 121 | 116 | 127
umol/L
  Creatinine at Week 24 | -0.3 (20.40) | 1.2 (10.83) | 5.7 (10.64) | 1.4 (8.53)
  Direct bilirubin at Week 24 | -0.1 (0.79) | 0.1 (0.84) | -0.1 (1.17) | -0.1 (1.01)
  Total bilirubin at Week 24 | -0.1 (3.33) | -0.1 (2.82) | 0.0 (3.66) | -0.8 (3.89)

28. Secondary Outcome: Change From Baseline in Hematology Parameters Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, Segmented Neutrophils, Total Neutrophils, White Blood Cell Count at Week 24
Description: Hematology parameters included basophils, eosinophils, lymphocytes, monocytes, platelet count, segmented neutrophils, total neutrophils, white blood cell count. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: giga cells per liter
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 117 | 121 | 115 | 124
giga cells per liter
  Basophils at Week 24 | 0.001 (0.0168) | 0.002 (0.0189) | 0.003 (0.0183) | -0.001 (0.0173)
  Eosinophils at Week 24 | -0.011 (0.0923) | -0.006 (0.0858) | -0.004 (0.1272) | -0.004 (0.0997)
  Lymphocytes at Week 24 | -0.037 (0.4182) | -0.075 (0.4373) | -0.151 (0.3949) | -0.047 (0.5084)
  Monocytes at Week 24 | -0.002 (0.1415) | -0.007 (0.1403) | 0.000 (0.1643) | -0.008 (0.1306)
  Platelet count at Week 24: number analyzed (Participants) | 117 | 119 | 115 | 123
  Platelet count at Week 24 | -4.8 (33.13) | -8.7 (32.33) | -5.3 (36.83) | -9.4 (36.13)
  Segmented neutrophils at Week 24 | 0.002 (1.2619) | 0.015 (1.3909) | 0.163 (1.2329) | -0.109 (1.1543)
  Total neutrophils at Week 24 | 0.002 (1.2619) | 0.015 (1.3909) | 0.163 (1.2329) | -0.110 (1.1550)
  White blood cell count at Week 24 | -0.05 (1.357) | -0.08 (1.551) | 0.01 (1.295) | -0.17 (1.288)

29. Secondary Outcome: Change From Baseline in Hematology Parameter Hematocrit
Description: Hematology parameter included hematocrit. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 118 | 122 | 116 | 124
Ratio | 0.0038 (0.02264) | 0.0037 (0.02242) | -0.0003 (0.02509) | 0.0002 (0.02351)

30. Secondary Outcome: Change From Baseline in Hematology Parameters Hemoglobin and Mean Corpuscle Hemoglobin Concentration at Week 24
Description: Hematology parameter included hemoglobin and mean corpuscle hemoglobin concentration. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 145 | 145 | 133 | 151
grams per liter
  Hemoglobin at Week 24: number analyzed (Participants) | 118 | 122 | 116 | 124
  Hemoglobin at Week 24 | -1.1 (7.24) | -1.6 (7.40) | -1.8 (8.06) | -1.6 (7.55)
  Mean corpuscle hemoglobin concentration at Week 24: number analyzed (Participants) | 114 | 117 | 113 | 122
  Mean corpuscle hemoglobin concentration at Week 24 | -5.3 (8.99) | -5.9 (9.74) | -3.9 (9.73) | -4.2 (9.64)

31. Secondary Outcome: Change From Baseline in Hematology Parameter Mean Corpuscle Hemoglobin at Week 24
Description: Hematology parameter included mean corpuscle hemoglobin. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 114 | 117 | 113 | 122
picograms | -0.21 (0.949) | -0.19 (1.173) | -0.10 (1.023) | -0.08 (0.830)

32. Secondary Outcome: Change From Baseline in Hematology Parameter Mean Corpuscle Volume and Mean Platelet Volume at Week 24
Description: Hematology parameter included mean corpuscle volume and mean platelet volume. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 145 | 145 | 133 | 151
femtoliters
  Mean corpuscle volume at Week 24: number analyzed (Participants) | 118 | 122 | 116 | 124
  Mean corpuscle volume at Week 24 | 0.8 (2.84) | 1.4 (2.45) | 0.6 (2.35) | 0.9 (2.43)
  Mean platelet volume at Week 24 | -0.01 (0.711) | -0.04 (0.626) | 0.13 (0.715) | 0.03 (0.627)

33. Secondary Outcome: Change From Baseline in Hematology Parameter Red Blood Cell Count at Week 24
Description: Hematology parameter included red blood cell count. Baseline was defined as the value at Visit 3 (Week 0). Change from Baseline was obtained by subtracting the Baseline value from the post-randomization value at Week 24.
Time Frame: Baseline (Week 0) and Week 24
Population: Safety population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: trillion cells per liter
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 114 | 117 | 113 | 122
trillion cells per liter | -0.03 (0.276) | 0.01 (0.256) | -0.08 (0.329) | -0.07 (0.262)

34. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings as Assessed by Investigator and Central Cardiologist
Description: The clinical interpretation of the ECG by the investigator was recorded as Normal, Abnormal but not clinically significant (ANCS) and Abnormal clinically significant (ACS). ECG interpretation by the central cardiologist included the most extreme result of the available ECGs where the central cardiologist's interpretation of the ECG was recorded as Normal, Unable to Evaluate and Abnormal. Data has been presented for number of participants with most severe on-treatment abnormal ECG findings.
Time Frame: Upto Week 24
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
Number analyzed (Participants) | 145 | 145 | 133 | 151
Participants
  Investigator interpretion ANCS: number analyzed (Participants) | 121 | 131 | 119 | 134
  Investigator interpretion ANCS | 58 | 60 | 59 | 67
  Investigator interpretion ACS: number analyzed (Participants) | 121 | 131 | 119 | 134
  Investigator interpretion ACS | 0 | 1 | 0 | 2
  Central cardiologist interpretation abnormal: number analyzed (Participants) | 120 | 131 | 119 | 136
  Central cardiologist interpretation abnormal | 49 | 51 | 51 | 59

35. Secondary Outcome: Exposure Estimates for SB-742457 Area Under Curve Over the Dosing Interval at Steady State (AUCτss)
Description: A total of five pharmacokinetic samples per participant were collected for the purpose of assessing plasma concentrations of SB-742457 and donepezil. At each visit (Day 28±5, 56±5, 84±5, 126±5 and 168±5) one sample was collected post 24 hours of last dose.
Time Frame: One sample at Day 28±5, 56±5, 84±5, 126±5 and 168±5 post 24 hours of last dose
Population: Pharmacokinetic concentration population comprised of all participants for whom a pharmacokinetic sample was obtained and analyzed. Only those participants with data available at the time of analysis were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hour per milliliter
Arm/Group | SB-742457-15mg | SB-742457-35mg
Number analyzed (Participants) | 141 | 132
nanograms hour per milliliter | 1434.89 (36.04) | 3424.91 (38.04)

36. Secondary Outcome: Exposure Estimates for SB-742457 Minimum Concentration at Steady State (Cmin-ss)
Description: Blood sample for pharmacokinetic analysis, were obtained within 24 hours of last dose. A total of five pharmacokinetic samples per participants were taken at Weeks 4, 8,12,18 and Week 24. The SB-742457 exposures at steady state Cmin-ss for each participant were estimated via nonlinear mixed effect analysis. Data has been presented in a consolidated format for SB-742457 exposures at steady state Cmin-ss.
Time Frame: One sample at Day 28±5, 56±5, 84±5, 126±5 and 168±5 post 24 hours of last dose
Population: Pharmacokinetic concentration population. Only those participants with data available at the time of analysis were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | SB-742457-15mg | SB-742457-35mg
Number analyzed (Participants) | 141 | 132
nanograms per milliliter | 46.03 (109.69) | 37.47 (39.47)

37. Secondary Outcome: Exposure Estimates for Donepezil Average Concentration at Steady State (Cavgss)
Description: Blood sample for pharmacokinetic analysis, were obtained within 24 hours of last dose. A total of five pharmacokinetic samples per participants were taken at Weeks 4, 8,12,18 and Week 24. The Donepezil exposures at steady state Cavgss for each participant were estimated via nonlinear mixed effect analysis. Data has been presented in a consolidated format for SB-742457 exposures at steady state Cavgss.
Time Frame: Weeks 4, 8,12,18 and Week 24
Population: as for outcome 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Groups:
- Donepezil 5 mg; Donepezil 10 mg: Participants received Donepezil capsule by one-step titration 5mg Donepezil once daily (Week 1 to Week 4) before up-titrating at Visit 4 (Week 4) to 10 mg once daily dose for the remaining 20 weeks of the treatment period (Week 4 to 24) along with matching placebo to SB-747457.
Arm/Group | Donepezil 5 mg | Donepezil 10 mg
Number analyzed (Participants) | 132 | 133
nanograms per milliliter | 17.53 (50.51) | 31.80 (60.14)

ADVERSE EVENTS:
Time Frame: Upto Week 24.
Description: Safety population was used for analysis.
Arm/Group | Placebo | SB-742457-15mg | SB-742457-35mg | Donepezil
All-Cause Mortality (participants affected / at risk) | 1/145 | 0/145 | 1/133 | 1/151
Serious Adverse Events (participants affected / at risk) | 7/145 | 7/145 | 3/133 | 10/151
Other Adverse Events (participants affected / at risk) | 42/145 | 39/145 | 38/133 | 62/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | SB-742457-15mg (N=145) | SB-742457-35mg (N=133) | Donepezil (N=151)
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ear injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | SB-742457-15mg (N=145) | SB-742457-35mg (N=133) | Donepezil (N=151)
Nasopharyngitis (Infections and infestations) | 3 | 3 | 3 | 4
Influenza (Infections and infestations) | 2 | 2 | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 4 | 3 | 3
Bronchitis (Infections and infestations) | 2 | 3 | 1 | 1
Cystitis (Infections and infestations) | 0 | 1 | 1 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 2
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 5 | 2 | 5
Dizziness (Nervous system disorders) | 1 | 3 | 2 | 5
Syncope (Nervous system disorders) | 1 | 1 | 1 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1
Clonus (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 5
Agitation (Psychiatric disorders) | 0 | 1 | 2 | 0
Hallucination (Psychiatric disorders) | 2 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 3
Sleep disorder (Psychiatric disorders) | 1 | 0 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Delusion of replacement (Psychiatric disorders) | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 1
Libido increased (Psychiatric disorders) | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 2
Application site rash (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 4
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Red blood cells urine (Investigations) | 0 | 0 | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 2 | 0 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Retinal infarction (Eye disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.